CLINICAL TRIAL: NCT06676358
Title: Evaluation of the Effects of Smoking on Trabecular Bone Microarchitecture Using CBCT in Periodontal Disease
Status: Completed | Type: Observational
Sponsor: Okan University (Other)
Responsible Party: Principal Investigator, Sibel Kayaalti-Yuksek, Assoc.Prof, Okan University
Other Study IDs: 2024/178-23; 2024/178-23 (Registry Identifier: ISTANBUL OKAN UNIVERSITY)
Record Dates: First submitted 2024-11-03; First posted 2024-11-06 (Actual); Last update posted 2024-11-06 (Actual); Status verified 2024-11

CONDITIONS: Cone Beam Computed Tomography; Periodontitis; Diagnosis of Bone Quality; Diagnosis, Oral; Smoking, Cigarette
Keywords: cone beam computed tomography; Periodontitis; Diagnosis
MeSH Terms: conditions — Periodontitis; Disease; Cigarette Smoking

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (6):
- Group 1: Non-Smokers with gingivitis: Patients with no history of cigarette use were assigned to the non-smoking group. Gingivitis was diagnosed based on the presence of bleeding on probing in at least 10% of all assessed sites and the absence of attachment and bone loss.
- Group 2: Smokers with gingivitis: Smoking status was categorized as follows: patients in the smoking group were those who smoked more than ten cigarettes daily and had a smoking history exceeding five years. Gingivitis was diagnosed based on the presence of bleeding on probing in at least 10% of all assessed sites and the absence of attachment and bone loss.
- Group 3: Smokers with mild moderate periodontitis: Smoking status was categorized as follows: patients in the smoking group were those who smoked more than ten cigarettes daily and had a smoking history exceeding five years. The classification of periodontitis stages was primarily based on clinical attachment loss (CAL), radiographic bone loss, and tooth loss criteria. Specifically, CAL of 1-2 mm was classified as periodontitis stage I, 3-4 mm as stage II (mild moderate periodontitis.)
- Group 4: Non-Smokers with mild moderate periodontitis: Patients with no history of cigarette use were assigned to the non-smoking group. The classification of periodontitis stages was primarily based on clinical attachment loss (CAL). Specifically, CAL of 1-2 mm was classified as stage I, 3-4 mm as stage II (mild moderate periodontitis).
- Group 5: Smokers with severe periodontitis: Smoking status was categorized as follows: patients in the smoking group were those who smoked more than ten cigarettes daily and had a smoking history exceeding five years. Clinical attachment loss of 1-2 mm was classified as and ≥5 mm as stages III-IV. The criteria for tooth loss included up to four teeth lost for stage III, and five or more teeth lost due to periodontitis for stage IV (severe periodontitis)
- Group 6: Non-Smokers with severe periodontitis: Patients with no history of cigarette use were assigned to the non-smoking group. Clinical attachment loss of 1-2 mm was classified as and ≥5 mm as stages III-IV. The criteria for tooth loss included up to four teeth lost for stage III, and five or more teeth lost due to periodontitis for stage IV (severe periodontitis)

SUMMARY:
The purpose of this cross-sectional study is to evaluate the morphometric properties of trabecular bone quality using Cone-beam computed tomography in periodontal disease at different stages, comparing smokers and non-smokers.

DETAILED DESCRIPTION:
This cross-sectional study aimed to analyze changes in trabecular bone quality associated with smoking inindividuals with periodontal disease using morphometric analysis of Cone Beam Computed Tomography (CBCT)images. Materials-Methods: The study involved 90 systemically healthy patients who were smokers (>=10cigarettes/day) or non-smokers, and were indicated for CBCT.Clinical periodontal parameters (plaque index, gingival index, probing pocket depth, bleeding on probing, clinicalattachment loss (CAL)) were recorded. Participants were divided into two main groups based on smoking statusand three subgroups based on periodontal diagnosis: gingivitis, Stage I-II periodontitis, and Stage III-IVperiodontitis (n=15). Mandibular first molars and central incisors without prosthetic restorations, endodonticlesions, or root canal treatments were included. Two volumetric regions of interest (ROIs) with dimensions of5x5x10 mm were selected around the apices of these teeth: posterior ROI and anterior ROI. Trabecular bonemicro-architecture was analyzed using the BoneJ plugin for morphometric parameters: anisotropy (DA), bonevolume fraction (BV/TV), trabecular thickness (Tb.Th), and trabecular separation (Tb.Sp). Statistical analysis wasperformed using Student's t-test, one-way ANOVA, and Kruskal-Wallis tests.

ELIGIBILITY:
Inclusion Criteria:

* Individuals aged 18 years or older who are systemically healthy.
* Presence of mandibular molars and mandibular anterior teeth.
* No pathologies affecting the alveolar bone.
* No history of orthodontic treatment.
* No use of medication that may impact bone health.
* No history of radiation or chemotherapy treatment.
* Selected mandibular molars and central incisors must be free of caries. Selected teeth must not have crowns, root canal treatments, or endodontic lesions.

Exclusion Criteria:

* Patients who are exhibiting signs of occlusal trauma
* Patients who are bruxism

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: A sample size of 15 patients per group (6 groups, total 90 patients) was calculated using the G*Power 3.1.9.2 software (power [1-β] = 0.80, alpha level [α] = 0.05, effect size [f] = 0.4)
Sampling Method: Non-Probability Sample
Enrollment: 90 (Actual)
Dates: Start 2024-03-15 (Actual); Primary Completion 2024-10-14 (Actual); Study Completion 2024-10-30 (Actual)

PRIMARY OUTCOMES:
Bone morphometric parameters | Baseline
  The microarchitecture of trabecular bone was analyzed by measuring bone morphometric parameters (BMPs) using the BoneJ plugin of the software.
  Degree of Anisotropy (DA): This parameter assesses the directional characteristics of trabecular bone. A DA value of 1 indicates an isotropic structure, while values above 1 indicate anisotropy. DA is calculated as the ratio of the longest mean intercept length vector to the shortest.
Bone morphometric parameters | Baseline
  Bone Volume Fraction (BV/TV): Representing the ratio of bone volume to total volume within the ROI, BV/TV indicates bone density.
Bone morphometric parameters | Baseline
  Trabecular Separation (Tb.Sp): Representing the mean distance between adjacent trabeculae, this parameter is also assessed using three-dimensional techniques.
Bone morphometric parameters | Baseline
  Trabecular Thickness (Tb.Th): This parameter indicates the average thickness of the trabeculae, obtained through direct three-dimensional assessment methods.

SECONDARY OUTCOMES:
Clinical periodontal parameters | Baseline
  A single calibrated operator (I.C.) performed the periodontal assessment utilizing an intraoral mirror and William's periodontal probe. Plaque Index (PI): The PI assesses the thickness of plaque along the gingival margin. After drying the teeth, the examiner visually inspects the surfaces of the teeth. Scores are assigned based on the presence and thickness of plaque on the gingival third of the tooth surface, usually on a scale from 0 (no plaque) to 3 (abundant plaque accumulation).
Clinical periodontal parameters | Baseline
  Gingival Index (GI): The GI measures the severity of gingival inflammation. The gingiva around selected teeth is observed and gently probed to evaluate bleeding and inflammation. Scores range from 0 to 3, where 0 indicates healthy gingiva and 3 indicates severe inflammation with spontaneous bleeding.
Clinical periodontal parameters | Baseline
  Periodontal Pocket Depth (PPD): PPD is measured by inserting a periodontal probe, like a William's probe, into the sulcus or pocket between the tooth and gum. The depth, in millimeters, is recorded for each probing site around the tooth to evaluate the extent of pocketing or detachment of the gingiva.
Clinical periodontal parameters | Baseline
  Clinical Attachment Level (CAL): CAL assesses the extent of periodontal attachment loss. It's measured as the distance from the cemento-enamel junction (CEJ) to the base of the pocket or sulcus. By comparing this measurement over time, one can evaluate the progression of periodontal disease.
Clinical periodontal parameters | Baseline
  Bleeding on Probing (BOP): BOP evaluates the presence of inflammation through bleeding. After probing the periodontal pocket, the site is observed for bleeding

CONTACTS AND LOCATIONS:
Locations (1):
- Okan Univercity, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kayaalti Yuksek S, Buyuk C, Cebeci I, Cayir Keles G. Evaluation of the Effects of Smoking on Trabecular Bone Microarchitecture Using Cone-Beam Computed Tomography in Periodontal Disease. Cureus. 2025 Dec 9;17(12):e98851. doi: 10.7759/cureus.98851. eCollection 2025 Dec. PMID 41523571